CLINICAL TRIAL: NCT03235167
Title: Cytidine-phosphate-guanosine (CpG) DNA in Hepatocellular Carcinoma Combination Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dalian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: zsyy_zxsys2017-07
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CpG DNA (Experimental): CpG DNA concentrate
  Interventions: Drug: CpG DNA; Procedure: transcatheter arterial chemoembolization
- placebo (Placebo Comparator): placebo concentrate
  Interventions: Procedure: transcatheter arterial chemoembolization; Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: CpG DNA — CpG DNA concentrate
  Arms: CpG DNA
Procedure: transcatheter arterial chemoembolization — transcatheter arterial chemoembolization (TACE) therapy for liver cancer
Drug: Placebo - Concentrate — CpG DNA vehicle
  Arms: placebo

SUMMARY:
to observe the outcome of hepatocellular carcinoma patients under the combination treatment of transcatheter arterial chemoembolization (TACE) and CpG DNA

ELIGIBILITY:
Inclusion Criteria:

* TNM (tumor node metastasis ) staging with non distant metastasis; no other tumors

Exclusion Criteria:

* having received previous treatment for liver cancer

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
survival time | 5 years
metastasis free survival time | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: xiaolin Yuan, Principal Investigator — Affiliated Zhongshan Hospital of Dalian University

IPD SHARING:
Plan to Share IPD: Undecided
age, gender, cancer staging